CLINICAL TRIAL: NCT03648489
Title: An International Multi-centre Randomised Phase II Study to Assess the Efficacy of TAK228 in Combination With Intravenous Weekly Paclitaxel Compared With Weekly Paclitaxel Alone in Women With Advanced/Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer (of Clear Cell, Endometrioid and High Grade Serous Type, and Carcinosarcoma)
Brief Title: Dual mTorc Inhibition in advanCed/Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer (of Clear Cell, Endometrioid and High Grade Serous Type, and Carcinosarcoma)
Acronym: DICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry); North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C/30/2011
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinosarcoma; Ovarian Serous Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Clear Cell Adenocarcinoma; Fallopian Tube Cancer; Fallopian Tube Neoplasms; Primary Peritoneal Carcinoma; Primary Peritoneal Serous Adenocarcinoma
Keywords: TAK228; TAK-228; Paclitaxel; Ovarian cancer; Platinum resistant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Weekly paclitaxel alone (Active Comparator): Paclitaxel, concentrate for solution for infusion 80mg per metre squared on day 1, 8 and 15 of a 28 day cycle. Cycles continue until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria
  Interventions: Drug: Paclitaxel
- Arm 2: Weekly paclitaxel plus TAK228 (Experimental): Paclitaxel, concentrate for solution for infusion 80mg per metre squared on day 1, 8 and 15 of a 28 day cycle. Cycles continue until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria
  TAK228, oral capsule 4mg on days 2-4, 9-11, 16-18 and 23-25 of a 28 day cycle i.e. in concurrence with paclitaxel. Cycles continue until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria
  Interventions: Drug: Paclitaxel; Drug: TAK228

INTERVENTIONS:
Drug: Paclitaxel — Please refer to arm/group description
Drug: TAK228 — Please refer to arm/group description
  Arms: Arm 2: Weekly paclitaxel plus TAK228

SUMMARY:
DICE is a randomised study recruiting 126 women over 3 years from hospitals in the UK and Germany. Eligible patients will have tissue based diagnosis of advanced/recurrent ovarian cancer (clear cell, endometrioid or high grade serous or carcinosarcoma), have had chemotherapy before, and be platinum-resistant (the cancer has returned/grown significantly during or within 6 months of platinum-containing chemotherapy).

DETAILED DESCRIPTION:
This study is for women with ovarian cancer that has come back following treatment, and is resistant to platinum chemotherapy. Weekly paclitaxel chemotherapy is standard for these women, but there is a need to provide more effective treatments. TAK228 is an unlicensed oral drug that blocks the PI3K/AKT/mTOR pathway, which is important to the survival and spread of cancer cells. When TAK228 is combined with paclitaxel in the laboratory, the anti-cancer effect of both is increased. The DICE trial will show whether using TAK228 in combination with weekly paclitaxel is more effective at treating the patient population than weekly paclitaxel alone. DICE will also look for 'biomarkers' that measure the activity of the cancer and the effects of treatment. This may help us understand which women might benefit from receiving TAK228 and weekly paclitaxel in future.

Randomisation will be to one of 2 groups (63 women in each). Treatment is divided into 4 week 'cycles':

Group 1: weekly paclitaxel for 3 weeks followed by 1 week rest each cycle

Group 2: weekly paclitaxel (see Group 1) plus TAK228 for 12 days each cycle

Women will stop treatment when the cancer grows significantly, there are unacceptable side effects, or the investigator and/or patient decides to stop. Women will be followed up until 6 months after the last patient receiving study treatment stops that treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent prior to admission to the study and initiation of any study procedures in accordance with ICH-GCP guidelines and to the local legislation
* Females ≥ 18 years of age
* Pathological diagnosis of ovarian, fallopian tube or primary peritoneal cancer, of clear cell, endometrioid or high grade serous subtype or carcinosarcoma. Local tumour board/MDT histological review is required and in mixed tumours more than 50% endometrioid, clear cell or high grade serous elements are required to define the predominant histology
* Platinum-resistant (recurrence within 6 months of platinum treatment), or platinum refractory disease (recurrence during platinum treatment), patients having received at least one prior line of chemotherapy. Carboplatin and weekly paclitaxel are permitted as first line therapy and/or as therapy for recurrent platinum sensitive disease i.e. prior to platinum resistant relapse
* Measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 by CT or MRI
* Fresh tumour biopsy during screening is compulsory if judged technically feasible by radiologist, unless the local site is unable to collect the sample due to COVID-19 capacity restrictions
* Patients with a history of brain metastasis are eligible as long as all the following criteria are met: brain metastases must have been treated, have no evidence of progression or haemorrhage after treatment, have been off dexamethasone for 4 weeks prior to first study treatment, and no ongoing requirement for dexamethasone or anti-epileptic drugs
* Available blocks for immunohistochemistry (IHC) and tissue microarray (TMA) or, if no block is available, 20 ordinary unstained slides (5µm sections) will be acceptable
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Adequate organ and bone marrow function
* Female patients who are postmenopausal for ≥ 1 year before the screening visit OR are surgically sterile OR if of childbearing potential, patient agrees to practice 1 highly effective and 1 additional effective method of contraception or true abstinence from informed consent to 90 days after the last dose of study treatment
* For women of child-bearing potential, negative blood serum pregnancy test within 14 days prior to the first study treatment
* Able to swallow oral medication

Exclusion Criteria:

* Previous treatment with PI3K, AKT, dual PI3K/mTOR inhibitors, mTORC1/2 inhibitors or mTORC1 inhibitors
* Prior weekly single agent paclitaxel
* Known allergy to paclitaxel and/or any excipients of investigational medicinal products that, in the investigator's opinion, precludes study treatment on clinical and/or safety grounds
* Treatment with strong inhibitor/s and/or inducer/s of cytochrome P450 (CYP) 3A4 or CYP2C8 within 7 days of study treatment
* Central nervous system (CNS) metastasis, for patients who have brain metastases, they will be eligible if their brain metastases must have been treated, have no evidence of progression or haemorrhage after treatment, have been off dexamethasone for 4 weeks prior to first study drug administration, and no ongoing requirement for dexamethasone or anti-epileptic drugs
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study
* Known human immunodeficiency virus infection
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* German sites only: Unable to be regularly followed up for any reason (geographic, familiar, social, psychological, housed in an institution e.g. prison because of a court agreement or administrative order)
* German sites only: Subjects that are dependent on the sponsor (and/or contracted body e.g. CRO) or investigational site as well as on the investigator
* Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study treatment, or previously diagnosed with another malignancy and evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Breast feeding or pregnant
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of TAK228. In addition, patients with enteric small bowel stomata are also excluded
* Treatment with any investigational products, chemotherapy or radiotherapy within 28 days, or major surgery within 21 days of study treatment
* History of any of the following within the last 6 months before administration of the first dose of study treatment:

  1. Ischemic myocardial event, including angina requiring therapy and artery revascularisation procedures
  2. Ischemic cerebrovascular event, including transient ischemic attack and artery revascularisation procedures
  3. Requirement for inotropic support (excluding digoxin) or serious (uncontrolled) cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation or ventricular tachycardia)
  4. Placement of a pacemaker for control of rhythm
  5. New York Heart Association (NYHA) Class III or IV heart failure
  6. Pulmonary embolism
* Significant active cardiovascular or pulmonary disease including:

  1. Uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg). Use of anti-hypertensive agents to control hypertension before first dose of study treatment is allowed.
  2. Pulmonary hypertension
  3. Uncontrolled asthma or O2 saturation < 90% by arterial blood gas analysis or pulse oximetry on room air
  4. Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention, or history of valve replacement
  5. Medically significant (symptomatic) bradycardia
  6. History of arrhythmia requiring an implantable cardiac defibrillator
  7. Baseline prolongation of the rate-corrected QT interval (QTc) e.g. repeated demonstration of QTc interval > 480 milliseconds, or history of congenital long QT syndrome, or additional risk factors for torsades de pointes (e.g. hypokalaemia, family history of long QT syndrome) and patients who use concomitant medications that prolong the QT/QTc interval
* Patients receiving systemic corticosteroids (either IV or oral steroids, excluding inhalers or low-dose hormone replacement therapy) within 1 week before administration of the first dose of study treatment
* Daily or chronic use of a proton pump inhibitor (PPI) and/or having taken a PPI within 7 days before receiving the first dose of study treatment
* Poorly controlled diabetes mellitus defined as glycosylated haemoglobin (HbA1c) > 7%; patients with a history of transient glucose intolerance due to corticosteroid administration may be enrolled in this study if all other inclusion/exclusion criteria are met

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS (as assessed by RECIST v1.1), defined as time from study entry to first evidence of disease progression or death due to any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) at 24 weeks | 6 months
  PFS (as assessed by RECIST v1.1) at 24 weeks, defined as time from study entry to first evidence of disease progression or death due to any cause
Overall Response Rate (ORR) | 12 months
  ORR (as assessed by RECIST v1.1) defined by complete response (CR) or partial response (PR)
Duration of Response (DOR) | 12 months
  DOR defined as time from study entry to change in response from CR or PR to stable disease (SD) or progressive disease (PD) (as assessed by RECIST v1.1)
Time to Progression (TTP) | 12 months
  TTP defined as time from study entry to first evidence of disease progression or death due to any cause
Clinical Benefit Rate (CBR) at 4 months | 4 months
  TTP defined as time from study entry to first evidence of disease progression or death due to any cause
Response according to Gynecologic Cancer Intergroup (GCIG) CA125 criteria | 12 months
  A response according to CA125 has occurred if there is at least a 50% reduction in CA125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 28 days. Patients can be evaluated according to CA125 only if they have a pretreatment sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment
Overall Survival (OS) | 12 months
  OS defined as time from study entry to death due to any cause or to study termination
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 12 months
  The number of patients experiencing 1 or more AEs will be summarised by the event name, relationship to study treatment and severity
Change from baseline quality of life (QOL) as assessed by EORTC QLQ-C30 questionnaire Global Health Status Domain | 12 months
  EORTC QLQ-C30 is used to assess the overall quality of life in cancer patients. It consists of 30 questions and 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status/QOL scale is scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in QOL or functioning and positive values indicate improvement
Change from baseline QOL as assessed by EORTC QLQ-OV28 questionnaire | 12 months
  EORTC QLQ-OV28 is used to assess the overall health-related quality of life in patients with local or advanced ovarian cancer. EORTC QLQ-OV28 consists of 28 questions evaluated across eight multi-item and 4 single item scales: abdominal/GI symptoms, peripheral neuropathy, hormonal symptoms, body image, attitude to disease/treatment, chemotherapy side effects, and sexuality, and single items scales for indigestion/heartburn, hair loss, upset due to hair loss, and taste. Questions use a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krell, Principal Investigator — Imperial College London
Locations (15):
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - KEM Kliniken Essen-Mitte, Essen
- United Kingdom (12):
  - Furness General Hospital, Barrow in Furness, Cumbria
  - St George's University Hospitals NHS Foundation Trust, London, Greater London
  - The Royal Marsden NHS Foundation Trust, London, Greater London
  - Imperial College Healthcare NHS Trust, London, Greater London
  - The Royal Marsden NHS Foundation Trust, Sutton, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Royal Lancaster Infirmary, Lancaster, Lancashire
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fiorentino F, Krell J, de la Rosa CN, Webber L. DICE: Dual mTorc Inhibition in advanCed/recurrent Epithelial ovarian cancer resistant to standard treatment-a study protocol for a randomised trial investigating a novel therapy called TAK228. Trials. 2022 Apr 5;23(1):261. doi: 10.1186/s13063-022-06201-3. PMID 35382842
- [Derived] de la Rosa CN, Krell J, Day E, Clarke A, Reddi M, Webber L, Fiorentino F. Statistical analysis plan for the Dual mTorc Inhibition in advanCed/recurrent Epithelial ovarian, fallopian tube or primary peritoneal cancer (of clear cell, endometrioid and high-grade serous type, and carcinosarcoma) trial (DICE). Trials. 2022 Jan 5;23(1):13. doi: 10.1186/s13063-021-05669-9. PMID 34986897